CLINICAL TRIAL: NCT01980472
Title: Phase II Trial of Geriatric Evaluation as Selection Criteria and Predictive Factor of Safety in Elderly Patients (≥ 70 Years) With Non-small Cell Lung Cancer (NSCLC)That Can be Treated With Bevacizumab, Carboplatin and Paclitaxel
Brief Title: Chemotherapy Plus Bevacizumab in Elderly Non-small Cell Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo de Investigación y Divulgación Oncológica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GIDO1201
Record Dates: First submitted 2013-10-14; First posted 2013-11-11 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Chemotherapy Regimen Plus Bevacizumab
Oversight: Data Monitoring Committee: No

ARMS (1):
- bevacizumab, carboplatin and paclitaxel (Experimental): bevacizumab, carboplatin and paclitaxel
  Interventions: Biological: bevacizumab, carboplatin and paclitaxel

INTERVENTIONS:
Biological: bevacizumab, carboplatin and paclitaxel — 4-6 initial cycles of bevacizumab, carboplatin and paclitaxel bevacizumab until progression or toxicity

SUMMARY:
A phase II Study of an adapted chemotherapy regimen plus bevacizumab in elderly non-small cell lung cancer patients selected by geriatric assessment

DETAILED DESCRIPTION:
CRITERIOS INCLUSION

* Written informed consent confirming that the patient understands the study objective and the procedures required.
* Patients must be able to accomplish with the study protocol.
* Men and women ≥70 years old.
* Histologically or cytologically confirmed diagnosis of non-squamous non-small cell lung cancer (NSCLC) with EGFR gen mutational status negative or non-determinable.
* Patients with stage IV disease.
* Patients who have not received first-line treatment
* Patients with ECOG performance status 0 or 1.
* Adequate bone marrow function, defined as:

  * Absolute neutrophil count (ANC) ≥1.500/mm3 or ≥1.5x109/L;
  * Hemoglobin ≥ 9 g/dL.
  * Platelet count ≥ 100.000/mm3.
* Adequate renal function, defined as:

  * Creatinine clearance ≥ 40 ml/min, according to MDRD formula.
  * Urine dipstick proteinuria <2+. If urine dipstick for proteinuria ≥2+ 24 hours urine must be collected within 24 hours, and proteins must be less than 1 g.
* Fertile males must use an effective contraceptive method (error rate per year <1%) during the trial and until 6 months after the last study treatment dose, such as sexual abstinence, previous vasectomy and/or having a partner using any of following methods: implantables, injections, combined oral contraceptives and/or intrauterine device (hormonal only).

CRITERIOS EXCLUSION

* Previous chemotherapy for advanced NSCLC.
* History of haemoptysis grade ≥ 2 (defined as at least 2.5 mL of bright red blood) in the 3 months before inclusion.
* Major surgery (including open biopsy), significant traumatic injuries in the 28 days before inclusion or anticipation of the need of major surgical procedure during the treatment period
* Minor surgery, including permanent catheter insertion, in the 24 hours before bevacizumab infusion.
* Untreated brain metastases. Patients with CNS metastases treated with radiotherapy or surgery may be included if there is no evidence of progression after treatment
* Radiological evidence of a tumor that invades or is adjacent to a main blood vessel (e.g. lung artery or superior cava venous).
* Radiotherapy, in any lesion and for any reason, within 28 days before inclusion. Palliative radiotherapy for bone lesions within 14 days before inclusion is allowed.
* Treatment with aspirin (>325 mg/day) or clopidogrel (>75 mg/day) within 10 days prior to bevacizumab first dose. Use of full dose of oral or parenteral anticoagulants or thrombolytic agents in therapeutic doses. Prophylactic use of anticoagulant therapy is allowed.
* Uncontrolled hypertension (systolic BP >140 mmHg, diastolic BP >90mmHg) in the 28 days previous to inclusion or history of hypertensive crisis, or hypertensive encephalopathy.
* Clinically significant cardiovascular disease (i.e. cerebrovascular accident (CVA), myocardial infarction within 6 months prior to inclusion, unstable angina, congestive cardiac insufficiency NYHA ≥ II, left ventricular ejection fraction (LVEF) <50% or serious cardiac arrhytmia), not responding to treatment or that can interfere with trial treatment administration.
* Not healed wounds, active peptic ulcer or untreated bone fracture.
* Hypersensibility to any of the active ingredients of the study treatment (bevacizumab, carboplatine and paclitaxel) or any of its excipients.
* Serious cognitive impairment that limits the patient to understand and answer the study questionnaires.
* Inability to comply with the study protocol and/or follow-up procedures due to psychological, familiar, social or geographical problems
* Patients with an ADL score <5 at the screening.
* Patients with dementia: 9-12 points in the Folstein MMS at the screening.
* Patients accomplishing fragility Balducci criteria at the screening:

  * Age ≥ 85 years old
  * Dependence in 1 or more ADL
  * >3 comorbilities
  * >1 geriatric syndrome

OBJETIVOS

To assess the toxicity of the treatment in elderly patients (≥70 years) with NSC lung cancer who meet inclusion criteria for bevacizumab and selected based on a geriatric evaluation.

Determine predictive factors of toxicity in the elderly population (≥70 years). Determine objective response rate Determine disease control rate Determine progression free survival Determine overall survival Determine safety of the treatment combination

VARIABLES

Primary endpoint:

Rate of grade 3-4 neutropenia defined according to National Cancer Institute Common Terminology Criteria version 4.0 (NCI-CTC v4.0).

Secondary endpoints:

* Items of the Comprehensive Geriatric Assessment (CGA) scale as predictive factors for toxicity end-points.
* Objective response according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1).
* Progression-free survival.
* Overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent confirming that the patient understands the study objective and the procedures required.
* Patients must be able to accomplish with the study protocol.
* Men and women ≥70 years old.
* Histologically or cytologically confirmed diagnosis of non-squamous non-small cell lung cancer (NSCLC) with EGFR gen mutational status negative or non-determinable.
* Patients with stage IV disease.
* Patients who have not received first-line treatment
* Patients with ECOG performance status 0 or 1.
* Adequate bone marrow function, defined as:

Absolute neutrophil count (ANC) ≥1.500/mm3 or ≥1.5x109/L; Hemoglobin ≥ 9 g/dL. Platelet count ≥ 100.000/mm3. • Adequate renal function, defined as: Creatinine clearance ≥ 40 ml/min, according to MDRD formula. Urine dipstick proteinuria <2+. If urine dipstick for proteinuria ≥2+ 24 hours urine must be collected within 24 hours, and proteins must be less than 1 g.

• Fertile males must use an effective contraceptive method (error rate per year <1%) during the trial and until 6 months after the last study treatment dose, such as sexual abstinence, previous vasectomy and/or having a partner using any of following methods: implantables, injections, combined oral contraceptives and/or intrauterine device (hormonal only).

Exclusion Criteria:

* Previous chemotherapy for advanced NSCLC.
* History of haemoptysis grade ≥ 2 (defined as at least 2.5 mL of bright red blood) in the 3 months before inclusion.
* Major surgery (including open biopsy), significant traumatic injuries in the 28 days before inclusion or anticipation of the need of major surgical procedure during the treatment period
* Minor surgery, including permanent catheter insertion, in the 24 hours before bevacizumab infusion.
* Untreated brain metastases. Patients with CNS metastases treated with radiotherapy or surgery may be included if there is no evidence of progression after treatment
* Radiological evidence of a tumor that invades or is adjacent to a main blood vessel (e.g. lung artery or superior cava venous).
* Radiotherapy, in any lesion and for any reason, within 28 days before inclusion. Palliative radiotherapy for bone lesions within 14 days before inclusion is allowed.
* Treatment with aspirin (>325 mg/day) or clopidogrel (>75 mg/day) within 10 days prior to bevacizumab first dose. Use of full dose of oral or parenteral anticoagulants or thrombolytic agents in therapeutic doses. Prophylactic use of anticoagulant therapy is allowed.
* Uncontrolled hypertension (systolic BP >140 mmHg, diastolic BP >90mmHg) in the 28 days previous to inclusion or history of hypertensive crisis , or hypertensive encephalopathy.
* Clinically significant cardiovascular disease (i.e. cerebrovascular accident (CVA), myocardial infarction within 6 months prior to inclusion, unstable angina, congestive cardiac insufficiency NYHA ≥ II, left ventricular ejection fraction (LVEF) <50% or serious cardiac arrhythmia), not responding to treatment or that can interfere with trial treatment administration.
* Not healed wounds, active peptic ulcer or untreated bone fracture.
* Hypersensibility to any of the active ingredients of the study treatment (bevacizumab, carboplatine and paclitaxel) or any of its excipients.
* Serious cognitive impairment that limits the patient to understand and answer the study questionnaires.
* Inability to comply with the study protocol and/or follow-up procedures due to psychological, familiar, social or geographical problems
* Patients with an ADL score <5 at the screening.
* Patients with dementia: 9-12 points in the Folstein MMS at the screening.
* Patients accomplishing fragility Balducci criteria at the screening:

Age ≥ 85 years old Dependence in 1 or more ADL >3 comorbidities >1 geriatric syndrome

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3-4 neutropenia defined according to National Cancer Institute Common Terminology Criteria version 4.0 (NCI-CTC v4.0) | participants will be followed for the duration of the study, around 3 years

SECONDARY OUTCOMES:
Plasma VEGF | participants will be followed for the duration of the study, around 3 years
Objective response and Stable disease according to RECIST | participants will be followed for the duration of the study, around 3 years
progression-free survival and overall survival | participants will be followed for the duration of the study, around 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Juan Vidal, Dr., Principal Investigator — Grup d'investigació i divulgació en oncologia
Locations (10):
- Spain (10):
  - Hospital Virgen de los Lirios, Alcoy, Valencia
  - Hospital de Castellón, Castellon, Valencia
  - Hospital de Elda, Elda, Valencia
  - Hospital de Manises, Manises, Valencia
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital San Juan, San Juan, Valencia
  - Hospital U. y P. La Fe, Valencia, Valencia
  - Hospital Lluis Alcanyis, Xátiva, Valencia
  - Hospital General de Alicante, Alicante
  - Hospital General de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: web of Sponsor — http://gido.es/